CLINICAL TRIAL: NCT00460928
Title: Preventive IVIG Therapy for Congenital Heart Block (The PITCH Study)
Brief Title: Preventive IVIG Therapy for Congenital Heart Block
Acronym: PITCH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Lupus Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-045
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Block; Neonatal Lupus; Autoantibody-associated Heart Block
Keywords: congenital heart block; neonatal lupus; systemic lupus erythematosus; Sjogren syndrome; autoantibodies; SSA/Ro; SSB/La; autoimmunity; pregnancy; intravenous immune globulin; IVIG; immunoglobulin
MeSH Terms: conditions — Congenital heart block; Neonatal Systemic lupus erythematosus; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Autoimmune Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- intravenous immune globulin (IVIG) (Experimental)
  Interventions: Drug: intravenous immune globulin (IVIG)

INTERVENTIONS:
Drug: intravenous immune globulin (IVIG)

SUMMARY:
Neonatal lupus (NL) is the name given to a group of conditions that can affect the babies of mothers who have certain autoantibodies against components of the body's cells that are called SSA/Ro and SSB/La. NL can appear as a temporary rash that usually goes away by the time the baby is 6 months old, or very rarely an abnormal blood or liver condition that also improves with time - or it can cause permanent and often life-threatening damage to the fetal heart, known as congenital heart block (CHB). In women with anti-Ro/La antibodies who are pregnant for the first time, only about 2% of the babies will develop CHB. But for a woman who has already had a child with CHB or NL rash, the risk of CHB in her next pregnancy is nearly 20%. Unfortunately, once complete (third degree) heart block has been unequivocally identified in a fetus, it has never been reversed with any of the therapies that have been tried to date. Our previous studies strongly indicate that scarring of the conduction system (the heart's own natural "pacemaker"), a consequence of inflammation triggered by the mother's antibodies, damages or even destroys the cells that allow the heart to beat at a normal rhythm. Instead, the damaged heart beats extremely slowly, to an extent that is fatal to nearly 20% of affected babies (with most deaths occurring as fetal demises). Nearly all surviving children with CHB require permanent implantation of a pacemaker device. Because it is so difficult to treat or repair the damaged heart, a high-priority strategy is to try to prevent the inflammatory process before irreversible scarring can occur. The aim of this clinical-based proposal is to determine whether treating the pregnant mother with intravenous immune globulin (IVIG) will prevent the development of CHB.

DETAILED DESCRIPTION:
Perhaps the strongest clinical association with autoantibodies against SSA/Ro-SSB/La is the development of congenital heart block (CHB) in an offspring, an alarming prospect facing 2% of primigravid mothers with these antibodies. Recurrence rates approach 20%. Disease can progress rapidly, with advanced block and life-threatening cardiomyopathy observed less than 2 weeks from normal sinus rhythm. Once 3rd degree (complete) block is identified, reversal has never been achieved, despite dexamethasone. This makes biologic sense since the signature lesion is fibrosis of the atrioventricular node. Thus, strategies aimed at preventing disease assume high priority. Although disease expression in the fetus requires additional factors to amplify the cascade to fibrosis, maternal anti-Ro/La antibodies are necessary. Accordingly, eliminating fetal exposure to these antibodies is a sound and important approach. Intravenous immune globulin (IVIG) is particularly exciting in its potential not only to lower maternal antibody levels (which is not accomplished with glucocorticoids or immunosuppression), but actually to influence effector mechanisms in the fetus itself. Aim 1 is a clinical trial to assess the efficacy of IVIG in preventing CHB. Proof of efficacy is challenging since CHB occurs in only 2% of first pregnancies of anti-Ro/La+ women. However, given the 10-fold higher risk of CHB in a pregnancy after the birth of child with neonatal lupus (NL), mothers with previous NL-affected children are the target population for study. Sample size calculations employ Simon's 2-stage optimal design. Based on a 2-sided significance level of 0.05, a power of 90% to show reduction of risk to 5% given the prediction that 18% of untreated subjects will get some degree of CHB, Stage 1 will enroll 19 women who have had a previous child with CHB or NL rash, to receive IVIG (400 mg/kg IVIG every 3 weeks for a total of 5 treatments) from weeks 12 through 24 of gestation. If fewer than 3 mothers have children with 2nd or 3rd degree block, then an additional 35 mothers will be enrolled in Stage 2 (total = 54 subjects). IVIG will be considered efficacious and worthy of further study if fewer than 6 of 54 subjects have a child with advanced CHB. Secondary outcomes include 1st degree block, myocardial injury absent conduction defects, and isolated endocardial fibroelastosis as assessed by serial fetal echocardiograms and EKG at birth.

Aim 2 will address: a) the effect of IVIG on antibody titer and subclass; b) genetic polymorphisms in Fc gamma receptor (FcgR) and platelet-activating factor acetylhydrolase and their potential association with response to IVIG; c) whether a decrease in anti-La antibodies positively correlates with the level of anti-La antiidiotypic antibodies; d) whether IVIG blocks expression of activation markers on human macrophages after challenge with opsonized apoptotic cardiocytes and whether this positively correlates with increased expression of the inhibitory Fc receptor, FcgRIIb.

In sum, IVIG is a promising agent that may have effects at several levels of the pathologic cascade to antibody-mediated CHB.

ELIGIBILITY:
Inclusion Criteria:

* Mother must currently have an intrauterine pregnancy of less than 12 weeks.
* Mother must have antibodies to SSA/Ro and/or SSB/La (will be confirmed in the clinical immunology laboratory at the Principal Investigator's institution, the NYU-Hospital for Joint Diseases).
* Mother can be asymptomatic or have any rheumatic disease (such as lupus, Sjogren syndrome or other).
* Mother must have had a previous child with one of the following: (a) congenital heart block (any degree) documented by EKG if live birth and/or echocardiogram if fetal demise; (b) characteristic neonatal lupus rash confirmed by photograph revealing annular lesions (evaluated by the PI), dermatology note, and/or biopsy; (c) congenital heart block and rash.
* Mother may be taking 20 mg prednisone per day or less.

Exclusion Criteria:

* Mother does not have antibodies to either SSA/Ro or SSB/La.
* Mother is taking greater than 20 mg prednisone per day.
* Mother has any condition that would contraindicate the use of IVIG: (a) prior serious reaction to IVIG infusion; (b) known IgA deficiency; (c) intolerance of volume load, e.g., congestive heart failure; (d) nephrotic syndrome.
* Identification in the fetus of any of the following structural lesions considered causal for congenital heart block: (a) atrioventricular septal defects; (b) single ventricle; (c) developmental tricuspid valve disease; (d) L-transposition of the great arteries; (e) heterotaxia.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
2nd or 3rd degree heart block | 1 Day

SECONDARY OUTCOMES:
Prolonged PR interval (>0.150 sec) | 1 Day
Sign of myocardial injury, w/o change in heart rate/rhythm | 1 Day
Echocardiographic density consistent with EFE | 1 Day
Fetal death | 1 Day
Rash consistent w neonatal lupus | 1 Day
Gestational age at birth | 1 Day
Birth weight | 1 Day
Abnormal fluid collection | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Buyon, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New York University School of Medicine / NYU-Hospital for Joint Diseases, New York, New York

REFERENCES:
- [Derived] Friedman DM, Llanos C, Izmirly PM, Brock B, Byron J, Copel J, Cummiskey K, Dooley MA, Foley J, Graves C, Hendershott C, Kates R, Komissarova EV, Miller M, Pare E, Phoon CK, Prosen T, Reisner D, Ruderman E, Samuels P, Yu JK, Kim MY, Buyon JP. Evaluation of fetuses in a study of intravenous immunoglobulin as preventive therapy for congenital heart block: Results of a multicenter, prospective, open-label clinical trial. Arthritis Rheum. 2010 Apr;62(4):1138-46. doi: 10.1002/art.27308. PMID 20391423
- See also: Evaluation of Fetuses in the Preventive IVIG Therapy for Congenital Heart Block (PITCH) study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3214993/?report=reader